CLINICAL TRIAL: NCT04820530
Title: A Multicenter, Single-arm, Open-label Trial to Evaluate Efficacy and Safety of Oral, Twice Daily Iptacopan in Adult PNH Patients Who Are Naive to Complement Inhibitor Therapy
Brief Title: Study of Efficacy and Safety of Twice Daily Oral Iptacopan (LNP023) in Adult PNH Patients Who Are Naive to Complement Inhibitor Therapy
Acronym: APPOINT-PNH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLNP023C12301; 2020-003172-41 (EudraCT Number)
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Results first posted 2023-11-15 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria (PNH)
Keywords: Paroxysmal nocturnal hemoglobinuria; Hemoglobin; Anemia; LNP023; Iptacopan
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal; Anemia | interventions — iptacopan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LNP023 (Experimental): Participants receive LNP023 at a dose of 200 mg orally b.i.d
  Interventions: Drug: Iptacopan (LNP023)

INTERVENTIONS:
Drug: Iptacopan (LNP023) — Taken orally b.i.d. Dosage supplied: 200mg Dosage form: Hard gelatin capsule Route of Administration: oral
  Other Names: Iptacopan

SUMMARY:
The purpose of this Phase 3 study was to determine whether iptacopan is efficacious and safe for the treatment of Paroxysmal nocturnal hemoglobinuria (PNH) patients who were naïve to complement inhibitor therapy.

DETAILED DESCRIPTION:
This study was a multicenter, single-arm, open-label trial which was comprised of 8 weeks screening period, 24-week core treatment period and 24-week extension treatment period.

Eligible PNH patients with hemolysis (LDH > 1.5 ULN) and anemia (hemoglobin <10 g/dL), who were naive to complement inhibitor therapy, including anti-C5 antibody treatment, received iptacopan monotherapy at a dose 200 mg orally b.i.d.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants ≥ 18 years of age with a diagnosis of PNH confirmed by high-sensitivity flow cytometry with RBCs and WBCs clone size ≥ 10%
* Mean hemoglobin level <10 g/dL
* LDH > 1.5 x Upper Limit of Normal (ULN)
* Vaccination against Neisseria meningitidis infection is required prior to the start of study treatment
* If not received previously, vaccination against Streptococcus pneumoniae and Haemophilus influenzae infections should be given

Exclusion Criteria:

* Prior treatment with a complement inhibitor, including anti-C5 antibody
* Known or suspected hereditary complement deficiency
* History of hematopoietic stem cell transplantation
* Patients with laboratory evidence of bone marrow failure (reticulocytes <100x109/L; platelets <30x109/L; neutrophils <0.5x109/L).
* Active systemic bacterial, viral (incl. COVID-19)or fungal infection within 14 days prior to study drug administration.
* History of recurrent invasive infections caused by encapsulated organisms, e.g. meningococcus or pneumococcus.
* Major concurrent comorbidities including but not limited to severe kidney disease (e.g., dialysis), advanced cardiac disease (e.g., NYHA class IV heart failure), severe pulmonary disease (e.g., severe pulmonary hypertension (WHO class IV)), or hepatic disease (e.g., active hepatitis) that in the opinion of the investigator precludes participant's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2023-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- China (2):
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Tianjin
- Novartis Investigative Site, Paris, France
- Germany (2):
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Essen
- Novartis Investigative Site, Avellino, AV, Italy
- Malaysia (2):
  - Novartis Investigative Site, Kota Kinabalu, Sabah
  - Novartis Investigative Site, Kuching, Sarawak
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, South Korea
- Novartis Investigative Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient level data and supporting clinical documents from eligible studies. these requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Derived] DeCastro C, Sheinberg P, Han B, Vallow S, Bermann G, Dhalke M, Kumar R, Dickie G, Galipeau N, Lamoureux R, Rupinski K, Lowe C, Nieves A, de Fontbrune FS, de Latour RP. Patient-Reported Meaningful Change in Symptoms and Impacts of Paroxysmal Nocturnal Hemoglobinuria (PNH) in Three Phase III Clinical Trials of Iptacopan. Patient. 2025 Nov;18(6):699-712. doi: 10.1007/s40271-025-00755-5. Epub 2025 Jul 22. PMID 40694294
- [Derived] Risitano AM, Kulasekararaj AG, Scheinberg P, Roth A, Han B, Maciejewski JP, Ueda Y, de Castro CM, Di Bona E, Fu R, Zhang L, Griffin M, Langemeijer SMC, Panse J, Schrezenmeier H, Barcellini W, Mauad VAQ, Schafhausen P, Tavitian S, Beggiato E, Chew LP, Gaya A, Huang WH, Jang JH, Kitawaki T, Kutlar A, Notaro R, Pullarkat V, Schubert J, Terriou L, Uchiyama M, Lee LWL, Yap ES, Frieri C, Marano L, de Fontbrune FS, Gandhi S, Trikha R, Alashkar F, Yang C, Liu H, Kelly RJ, Hochsmann B, Lawniczek T, Mahajan N, Solar-Yohay S, Kerloeguen C, Ferber P, Kumar R, Wang Z, Thorburn C, Maitra S, Li S, Verles A, Dahlke M, de Latour RP. Oral iptacopan monotherapy in paroxysmal nocturnal haemoglobinuria: final 48-week results from the open-label, randomised, phase 3 APPLY-PNH trial in anti-C5-treated patients and the open-label, single-arm, phase 3 APPOINT-PNH trial in patients previously untreated with complement inhibitors. Lancet Haematol. 2025 Jun;12(6):e414-e430. doi: 10.1016/S2352-3026(25)00081-X. PMID 40447351
- [Derived] Peffault de Latour R, Roth A, Kulasekararaj AG, Han B, Scheinberg P, Maciejewski JP, Ueda Y, de Castro CM, Di Bona E, Fu R, Zhang L, Griffin M, Langemeijer SMC, Panse J, Schrezenmeier H, Barcellini W, Mauad VAQ, Schafhausen P, Tavitian S, Beggiato E, Chew LP, Gaya A, Huang WH, Jang JH, Kitawaki T, Kutlar A, Notaro R, Pullarkat V, Schubert J, Terriou L, Uchiyama M, Wong Lee Lee L, Yap ES, Sicre de Fontbrune F, Marano L, Alashkar F, Gandhi S, Trikha R, Yang C, Liu H, Kelly RJ, Hochsmann B, Kerloeguen C, Banerjee P, Levitch R, Kumar R, Wang Z, Thorburn C, Maitra S, Li S, Verles A, Dahlke M, Risitano AM. Oral Iptacopan Monotherapy in Paroxysmal Nocturnal Hemoglobinuria. N Engl J Med. 2024 Mar 14;390(11):994-1008. doi: 10.1056/NEJMoa2308695. PMID 38477987
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 12 investigative sites in 8 countries: France(1), United Kingdom(1), Italy(1), Korea, Republic of(1), Singapore(1), China(3), Malaysia(2), Germany(2)
Pre-assignment Details: All patients provided written informed consent prior to the start of any study-related activities.
  Vaccination against Neisseria meningitidis, Streptococcus pneumoniae and Haemophilus influenzae infections was required prior to the start of treatment.
Groups:
- LNP023: Participants receive LNP023 at a dose of 200 mg b.i.d. orally
Period: Core Treatment Period
Arm/Group | LNP023
Started | 40
Completed | 40
Not Completed | 0
Period: Extension Treatment Period
Arm/Group | LNP023
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | LNP023
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (15.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 12
  Black or African American | 1
  Asian | 27

OUTCOME MEASURES:

1. Primary Outcome: Marginal Proportion (Expressed as Percentage) of Participants With Sustained Increase in Hemoglobin Levels From Baseline of ≥ 2 g/dL in the Absence of Red Blood Cell Transfusions
Description: Sustained increase in hemoglobin levels (responder) is defined as an increase from baseline in hemoglobin levels of ≥ 2 g/dL on three out of four measurements between Day 126 and 168 of the core treatment period, without requiring red blood cell (RBC) transfusions between Day 14 and Day 168. Requiring RBC transfusions refers to any patient receiving transfusions or meeting protocol defined criteria (Hemoglobin level of ≤9 g/dL (≤8 g/dL for Chinese population) with signs and or symptoms of sufficient severity to warrant a transfusion or Hemoglobin of ≤7 g/dL (≤6 g/dL for Chinese population), regardless of presence of clinical signs and/or symptoms).
  The term 'marginal proportion' can be interpreted as the population average probability of being a responder. Results incorporated a method to handle missing data using multiple imputation. Hence, all 40 patients enrolled contributed to the primary analysis.
Time Frame: Baseline, hemoglobin between Day 126 and Day 168 and absence of transfusions between Day 14 and Day 168
Population: Full Analysis Set (FAS): All patients with confirmed eligibility to whom study treatment was assigned.
Measure: Number (95% Confidence Interval); unit: Percentage of responders
Arm/Group | LNP023
Number analyzed (Participants) | 40
Percentage of responders | 92.2 [82.5 to 100.0]

2. Secondary Outcome: Marginal Proportion (Expressed as Percentage) With Sustained Hemoglobin Levels of ≥ 12 g/dL in the Absence of Red Blood Cell Transfusions
Description: Sustained hemoglobin levels (responder) is defined as hemoglobin levels ≥ 12 g/dL on three out of four measurements between Day 126 and 168 of the core treatment period, without requiring red blood cell (RBC) transfusions between Day 14 and Day 168. Requiring RBC transfusions refers to any patient receiving transfusions or meeting protocol defined criteria (Hemoglobin level of ≤9 g/dL (≤8 g/dL for Chinese population) with signs and or symptoms of sufficient severity to warrant a transfusion or Hemoglobin of ≤7 g/dL (≤6 g/dL for Chinese population), regardless of presence of clinical signs and/or symptoms).
  The term 'marginal proportion' can be interpreted as the population average probability of being a responder. Results incorporated a method to handle missing data using multiple imputation. Hence, all 40 patients enrolled contributed to the analysis.
Time Frame: Hemoglobin between Day 126 and Day 168 and absence of transfusions between Day 14 and Day 168
Population: Full Analysis Set (FAS): All patients with confirmed eligibility to whom study treatment was assigned.
Measure: Number (95% Confidence Interval); unit: Percentage of responders
Arm/Group | LNP023
Number analyzed (Participants) | 40
Percentage of responders | 62.8 [47.5 to 77.5]

3. Secondary Outcome: Marginal Proportion (Expressed as Percentage) of Participants Who Remain Free From Transfusions
Description: Marginal proportion (expressed as percentage) of participants who did not require transfusions between Day 14 and Day 168.
  Requiring RBC transfusions refers to any patient receiving transfusions or meeting protocol defined criteria (Hemoglobin level of ≤9 g/dL (≤8 g/dL for Chinese population) with signs and or symptoms of sufficient severity to warrant a transfusion or Hemoglobin of ≤7 g/dL (≤6 g/dL for Chinese population), regardless of presence of clinical signs and/or symptoms). The term 'marginal proportion' can be interpreted as the population average probability of being a responder.
  The 95% CI was obtained using the bootstrap method
Time Frame: Between Day 14 and Day 168
Population: Full Analysis Set (FAS): All patients with confirmed eligibility to whom study treatment was assigned.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LNP023
Number analyzed (Participants) | 40
Percentage of participants | 97.6 [92.5 to 100.0]

4. Secondary Outcome: Change From Baseline in Hemoglobin Levels in the Core Treatment Period
Description: Change from baseline in hemoglobin levels as mean of visits between Day 126 and Day 168.
  In order to factor out the effect of transfusions in this analysis, if a patient had a transfusion during the core treatment period, the hemoglobin (Hb) values during 30 days following the transfusion were excluded and Hb data were imputed.
  Change from baseline was analyzed using a mixed model of repeated measures which included age (indicator variable of age ≥ 45 years), sex, history of transfusion (yes/no) prior to study treatment, visit, and baseline hemoglobin as fixed effects and the interaction between visit and baseline hemoglobin levels.
Time Frame: Baseline, Day 126 to 168
Population: Full Analysis Set (FAS): All patients with confirmed eligibility to whom study treatment was assigned.
Measure: Mean (95% Confidence Interval); unit: g/dL
Arm/Group | LNP023
Number analyzed (Participants) | 40
g/dL | 4.28 [3.87 to 4.70]

5. Secondary Outcome: Percent Change From Baseline in LDH
Description: Percent change from baseline in lactate dehydrogenase (LDH) levels as mean of visits between Day 126 and Day 168.
  Percentage change from baseline was analyzed using a mixed model for repeated measures (MMRM) which includes age (indicator variable of age ≥ 45 years), sex, history of transfusion (yes/no) prior to study treatment, visit, baseline LDH as fixed effects and visit*baseline LDH as interaction.
  Results incorporated a method to handle missing data using multiple imputation. Hence, all 40 patients enrolled contributed to the analysis.
Time Frame: Baseline, Day 126 to 168
Population: Full Analysis Set (FAS): All patients with confirmed eligibility to whom study treatment was assigned.
Measure: Mean (95% Confidence Interval); unit: Percent change from baseline in LDH
Arm/Group | LNP023
Number analyzed (Participants) | 40
Percent change from baseline in LDH | -83.55 [-84.90 to -82.08]

6. Secondary Outcome: Adjusted Annualized Clinical BTH Rate in the Core Treatment Period
Description: Adjusted annualized rate of clinical breakthrough hemolysis (BTH) events is carried out using the Wilson method. The breakthrough is defined clinical if either there is a decrease in hemoglobin levels equal to or more than 2 g/dL (compared to the latest assessment, or within 15 days) or if patients present signs or symptoms of gross hemoglobinuria, painful crisis, dysphagia or any other significant clinical PNH-related signs & symptoms, in presence of laboratory evidence of intravascular hemolysis.
Time Frame: Between Day 1 and Day 168
Population: Full Analysis Set (FAS): All patients with confirmed eligibility to whom study treatment was assigned.
Measure: Number (95% Confidence Interval); unit: BTH events/year
Arm/Group | LNP023
Number analyzed (Participants) | 40
BTH events/year | 0.00 [0.00 to 0.17]

7. Secondary Outcome: Change From Baseline in Absolute Reticulocyte Count
Description: Change from baseline in absolute reticulocyte counts as mean of visits between Day 126 and Day 168.
  Change from baseline was analyzed using a MMRM which includes age (indicator variable of age ≥ 45 years), sex, history of transfusion (yes/no) prior to study treatment, visit, baseline reticulocyte counts as fixed effects and visit*baseline reticulocyte counts as interaction.
Time Frame: Baseline and mean of visits between Day 126 and 168
Population: Full Analysis Set (FAS): All patients with confirmed eligibility to whom study treatment was assigned.
Measure: Mean (95% Confidence Interval); unit: x10^9 cells/L
Arm/Group | LNP023
Number analyzed (Participants) | 40
x10^9 cells/L | -82.48 [-89.33 to -75.62]

8. Secondary Outcome: Change From Baseline in FACIT-Fatigue Score
Description: Change from baseline in FACIT-Fatigue scores as mean of visits between Day 126 and Day 168. The FACIT-Fatigue is a 13-item questionnaire with support for its validity and reliability in PNH that assesses patient self-reported fatigue and its impact on daily activities and function. All FACIT scales are scored so that a high score is better. As each of the 13 items of the FACIT-F Scale ranges from 0-4, the range of possible scores is 0-52, with 0 being the worst possible score and 52 the best.
  Change from baseline was analyzed using a Mixed Model of Repeated Measures (MMRM) which includes age (indicator variable of age ≥ 45 years), sex, history of transfusion (yes/no) prior to study treatment, visit, baseline FACIT-Fatigue score as fixed effects and visit*baseline FACIT-Fatigue score as interaction.
Time Frame: Baseline and mean of visits between Day 126 and Day 168
Population: Full Analysis Set (FAS): All patients with confirmed eligibility to whom study treatment was assigned.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | LNP023
Number analyzed (Participants) | 40
score on a scale | 10.75 [8.66 to 12.84]

9. Secondary Outcome: Adjusted Annualized Major Adverse Vascular Events Rate in the Core Treatment Period
Description: Adjusted annual rate is carried out using the Wilson method. A MAVE is defined as: acute peripheral vascular occlusion, amputation (non-traumatic; nondiabetic), cerebral arterial occlusion/cerebrovascular accident, cerebral venous occlusion, dermal thrombosis, gangrene (non-traumatic; nondiabetic), hepatic/portal vein thrombosis (Budd-Chiari syndrome), mesenteric/visceral arterial, thrombosis or infarction, mesenteric/visceral vein thrombosis or infarction, myocardial infarction, pulmonary embolus, renal arterial thrombosis, renal vein thrombosis, thrombophlebitis / deep vein thrombosis, transient ischemic attack, unstable angina or other.
Time Frame: Between Day 1 and Day 168
Population: Full Analysis Set (FAS): All patients with confirmed eligibility to whom study treatment was assigned.
Measure: Number (95% Confidence Interval); unit: MAVE events/year
Arm/Group | LNP023
Number analyzed (Participants) | 40
MAVE events/year | 0.00 [0.00 to 0.17]

10. Other Pre Specified Outcome: Percentage of Patients Meeting Hematological Response Criteria Irrespective of RBC Transfusions
Description: Patients with hematological response are those with an increase in Hb from baseline ≥ 2g/dL irrespective of red blood cell (RBC) transfusions and patients achieving Hb ≥ 12g/dL irrespective of RBC transfusions.
Time Frame: Baseline, Day 336
Population: Full analysis set: All patients with confirmed eligibility to whom study treatment was assigned. Only participants with valid Hb measurements at Day 336 were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | LNP023
Number analyzed (Participants) | 39
Percentage of participants
  ≥2 g/dL increase in Hb from baseline irrespective of RBC transfusions | 97.4
  Hb ≥ 12g/dL irrespective of transfusions | 79.5

11. Other Pre Specified Outcome: Marginal Proportion (Expressed as Percentage) of Patients Not Receiving and Not Requiring RBC Transfusions
Description: Requiring Red Blood Cells (RBC) transfusions refers to any patient receiving transfusions or meeting protocol defined criteria (Hemoglobin level of ≤9 g/dL (≤8 g/dL for Chinese population) with signs and or symptoms of sufficient severity to warrant a transfusion or Hemoglobin of ≤7 g/dL (≤6 g/dL for Chinese population), regardless of presence of clinical signs and/or symptoms).
Time Frame: Between Day 14 and Day 336
Population: Full analysis set: All patients with confirmed eligibility to whom study treatment was assigned.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LNP023
Number analyzed (Participants) | 40
Percentage of participants | 97.5 [92.5 to 100.0]

12. Other Pre Specified Outcome: Change From Baseline in Hemoglobin Levels
Description: Change from baseline in Hemoglobin at Visit Day 336
Time Frame: Baseline, Day 336
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | LNP023
Number analyzed (Participants) | 39
g/dL | 5.09 (2.010)

13. Other Pre Specified Outcome: Change From Baseline in LDH at Visit Day 336
Description: Change from baseline in Lactate dehydrogenase (LDH) at Visit Day 336
Time Frame: Baseline, Day 336
Population: Full Analysis Set (FAS): All patients with confirmed eligibility to whom study treatment was assigned.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | LNP023
Number analyzed (Participants) | 40
U/L | -1393.3 (652.15)

14. Other Pre Specified Outcome: Adjusted Annualized Clinical BTH Rate After the Start of LNP023 Treatment
Description: as for outcome 6
Time Frame: Between Day 1 and Day 336
Population: Full Analysis Set (FAS): All patients with confirmed eligibility to whom study treatment was assigned.
Measure: Number (95% Confidence Interval); unit: BTH events/year
Arm/Group | LNP023
Number analyzed (Participants) | 40
BTH events/year | 0.05 [0.01 to 0.17]

15. Other Pre Specified Outcome: Change From Baseline in Absolute Reticulocyte Count at Day 336
Description: Change from baseline in absolute reticulocyte count at visit Day 336.
Time Frame: Baseline, Day 336
Population: Full Analysis Set (FAS): All patients with confirmed eligibility to whom study treatment was assigned. Only participants with valid absolute reticulocyte count measurements at baseline and Day 336 were analyzed.
Measure: Mean (Standard Deviation); unit: x10^9 cells/L
Arm/Group | LNP023
Number analyzed (Participants) | 39
x10^9 cells/L | -76.55 (50.149)

16. Other Pre Specified Outcome: Change From Baseline in FACIT-Fatigue Score
Description: The FACIT-Fatigue is a 13-item questionnaire with support for its validity and reliability in PNH that assesses patient self-reported fatigue and its impact on daily activities and function. All FACIT scales are scored so that a high score is better. As each of the 13 items of the FACIT-F Scale ranges from 0-4, the range of possible scores is 0-52, with 0 being the worst possible score and 52 the best.
Time Frame: Baseline, Day 336
Population: Full Analysis Set (FAS): All patients with confirmed eligibility to whom study treatment was assigned. Only participants with valid FACIT-Fatigue scores at baseline and Day 336 were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LNP023
Number analyzed (Participants) | 39
score on a scale | 10.4 (10.14)

17. Other Pre Specified Outcome: Adjusted Annualized Major Adverse Vascular Events Rate After the Start of LNP023 Treatment
Description: Adjusted annual rate is carried out using the Wilson method. A Major Adverse Vascular Events (MAVE) is defined as: acute peripheral vascular occlusion, amputation (non-traumatic; nondiabetic), cerebral arterial occlusion/cerebrovascular accident, cerebral venous occlusion, dermal thrombosis, gangrene (non-traumatic; nondiabetic), hepatic/portal vein thrombosis (Budd-Chiari syndrome), mesenteric/visceral arterial, thrombosis or infarction, mesenteric/visceral vein thrombosis or infarction, myocardial infarction, pulmonary embolus, renal arterial thrombosis, renal vein thrombosis, thrombophlebitis / deep vein thrombosis, transient ischemic attack, unstable angina or other
Time Frame: Between Day 1 and Day 336
Population: Full Analysis Set (FAS): All patients with confirmed eligibility to whom study treatment was assigned.
Measure: Number (95% Confidence Interval); unit: MAVE events/year
Arm/Group | LNP023
Number analyzed (Participants) | 40
MAVE events/year | 0.00 [0.00 to 0.09]

ADVERSE EVENTS:
Time Frame: Adverse events of LNP023 group were reported from first dose of study treatment until the end of study treatment plus up to 30 days, up to a maximum duration of 48 weeks
Groups:
- LNP023 200mg b.i.d.: LNP023 200mg b.i.d.
Arm/Group | LNP023 200mg b.i.d.
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 8/40
Other Adverse Events (participants affected / at risk) | 24/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LNP023 200mg b.i.d. (N=40)
Breakthrough haemolysis (Blood and lymphatic system disorders) | 1
Cataract (Eye disorders) | 1
COVID-19 (Infections and infestations) | 2
Infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LNP023 200mg b.i.d. (N=40)
Abdominal pain (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 3
Pyrexia (General disorders) | 3
COVID-19 (Infections and infestations) | 7
Upper respiratory tract infection (Infections and infestations) | 7
Iron deficiency (Metabolism and nutrition disorders) | 3
Headache (Nervous system disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-03-28): https://cdn.clinicaltrials.gov/large-docs/30/NCT04820530/Prot_002.pdf
  • Statistical Analysis Plan (2022-11-17): https://cdn.clinicaltrials.gov/large-docs/30/NCT04820530/SAP_003.pdf